CLINICAL TRIAL: NCT00000179
Title: Agitation in Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: IA0003; 3U01AG010483-08S2 (NIH)
Record Dates: First submitted 1999-10-29; First posted 1999-11-01 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-03

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's disease; Psychomotor agitation; Behavioral symptoms; Haloperidol; Trazodone; Anti-psychotic agents; Anti-depressant agents
MeSH Terms: conditions — Alzheimer Disease; Psychomotor Agitation; Behavioral Symptoms | interventions — Trazodone; Haloperidol

INTERVENTIONS:
Drug: Trazodone
Drug: Haloperidol

SUMMARY:
Agitation affects 70 to 90 percent of patients with AD. Signs of agitation include verbal and physical aggressiveness, irritability, wandering, and restlessness. These behaviors often make caring for patients at home very difficult. Trazodone and haldol are two of the most commonly prescribed drugs for agitation in AD patients. Behavior management, a non drug approach, has been effective in reducing signs of agitation. Researchers have yet to compare the effectiveness of drug versus non drug therapy to treat agitation in AD patients and determine which is the best treatment. The Alzheimer's Disease Cooperative Study, with funding from the National Institute on Aging, is conducting an agitation treatment program at 21 sites in 16 States. This study will assess which of the above treatments is most effective.

ELIGIBILITY:
Inclusion Criteria:

* Memory problem consistent with a probable diagnosis of Alzheimer's disease (AD)
* Agitation symptoms for at least the past 2 weeks
* Patient has caregiver who can participate
* Patient lives in the same household as the caregiver

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Leon Thal, MD., Principal Investigator — University of California, San Diego
Locations (16):
- United States (16):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Southern Illinois University, Springfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - University of Massachusetts, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - New York University Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon

REFERENCES:
- [Result] Teri L, Logsdon RG, Peskind E, Raskind M, Weiner MF, Tractenberg RE, Foster NL, Schneider LS, Sano M, Whitehouse P, Tariot P, Mellow AM, Auchus AP, Grundman M, Thomas RG, Schafer K, Thal LJ; Alzheimer's Disease Cooperative Study. Treatment of agitation in AD: a randomized, placebo-controlled clinical trial. Neurology. 2000 Nov 14;55(9):1271-8. doi: 10.1212/wnl.55.9.1271. PMID 11087767
- See also: The Alzheimer's Disease Education and Referral (ADEAR) Center is a service of the National Institute on Aging (NIA) — http://www.alzheimers.org/